CLINICAL TRIAL: NCT00875199
Title: Contingency Management to Promote Weight Loss in Low Income Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UConn Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 09-108-2; 20090009 (Other Grant/Funding Number: The Ethel Donaghue Center for Translating Research into Practice and Policy)
Record Dates: First submitted 2009-03-31; First posted 2009-04-03 (Estimated); Last update posted 2011-11-21 (Estimated); Status verified 2011-11

CONDITIONS: Overweight
Keywords: Overweight; Obesity; Contingency Management
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Active Comparator): Participants assigned to Group A will receive the DPP manual (Wing & Gillis, 1996), a behavioral weight-loss program with demonstrated efficacy in facilitating weight loss. Participants in Group A will be instructed to read a section of the manual each week and complete suggested activities. They will also meet with the research staff once a week for weigh-in and supportive counseling.
  Interventions: Behavioral: weight loss manual-guided individual therapy sessions
- B (Experimental): Participants assigned to Group B will receive the DPP manual and will meet with research staff each week for weigh-in and supportive counseling. They will also receive contingency management or the opportunity to earn draws with the chance of winning prizes for losing weight and completing healthy activities.
  Interventions: Behavioral: contingency management

INTERVENTIONS:
Behavioral: contingency management — Prize-based contingency management for weight loss
  Arms: B
Behavioral: weight loss manual-guided individual therapy sessions — once weekly counseling session with research staff
  Arms: A

SUMMARY:
This study is designed to evaluate the feasibility and provide preliminary evidence for efficacy of a 12-week contingency management intervention to promote weight loss in overweight and obese low income adults in a community-based clinic. The study has three primary goals: (a) to determine if the contingency management treatment can be effectively applied to a new application, weight loss; (b) to obtain preliminary evidence for contingency management's efficacy in promoting weight loss and improving treatment retention, diet quality, physical activity levels, and self efficacy; and (c) to identify barriers and challenges to implementing contingency management for weight loss among low income patients.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 55 years
* body mass index in kg/m2 (BMI) between 25 and 39.9
* resting blood pressure between 90/60 and 140/90
* ability to speak English and read at the 6th grade level
* willingness to be randomly assigned to one of two groups

Exclusion Criteria:

* any serious acute or chronic medical problems that may impact dietary or exercise regimens
* psychiatric conditions

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2009-03; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
absolute and relative weight loss | pre-treatment, weekly during active phase, post-treatment
number of participants achieving clinically significant weight loss (5% or more of baseline weight) | pre-treatment, weekly during active phase, post-treatment

SECONDARY OUTCOMES:
retention | during active phase
changes on measures of diet quality, physical activity, and self-efficacy | pre-treatment, post-treatment
self-reports, focus groups | pre-treatment, post-treatment

CONTACTS AND LOCATIONS:
Overall Officials: Danielle M Barry, Ph.D., Principal Investigator — UConn Health
Locations (1):
- University of Connecticut Health Center, Farmington, Connecticut, United States